CLINICAL TRIAL: NCT07350785
Title: The Role of Monocyte Distribution Width (MDW) and Other Inflammatory Biomarkers in the Prediction of Mortality and Morbidity in Patients With Hip Fracture
Brief Title: Prediction of Mortality and Morbidity After Hip Fracture Using Monocyte Distribution Width (MDW)
Acronym: MDW
Status: Recruiting | Type: Observational
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, EFSTATHIOS CHRONOPOULOS, Professor in Orthopeadics at National and Kapodistrian University of Athens, Laboratory for Reasearch of the Musculoskeletal System Director, National and Kapodistrian University of Athens
Other Study IDs: 5570/04-03-2025
Record Dates: First submitted 2025-12-21; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Sepsis; Osteoporotic Hip Fracture; Hip Fracture
Keywords: Monocyte Distribution Width (MDW); Geriatric Patients; Inflammatory Biomarkers; Postoperative Mortality; Postoperative Morbidity; C-reactive Protein; Procalcitonin; Antithrombin III; Hip Fracture
MeSH Terms: conditions — Sepsis; Hip Fractures

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Peripheral venous blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Geriatric Patients With Hip Fracture: This cohort consists of patients aged 65 years or older who are admitted with a low-energy hip fracture and undergo surgical treatment. All participants receive standard-of-care clinical management according to institutional protocols. No experimental interventions are assigned as part of this study.
  Clinical data, medical history, and pre-fracture functional status are recorded at baseline. Blood samples are collected as part of routine care at hospital admission, postoperatively, and at discharge to measure complete blood count parameters, including Monocyte Distribution Width (MDW), and other inflammatory markers such as C-reactive protein, procalcitonin, and antithrombin III.
  Participants are followed postoperatively to assess clinical outcomes, including complications, morbidity, mortality, and health-related quality of life. Comparisons will be performed between subgroups defined by clinical outcomes or biomarker levels.

SUMMARY:
Hip fracture is a common injury in older adults and is often associated with serious complications, longer hospital stays, and increased risk of death. One of the most important causes of poor outcomes after hip fracture surgery is infection, including severe infections such as sepsis. Early identification of patients at higher risk for complications could help improve treatment and survival.

This study aims to examine whether a blood test parameter called Monocyte Distribution Width (MDW), along with other commonly used inflammatory markers, can help predict complications and survival in elderly patients with hip fracture. MDW is measured as part of a routine complete blood count and has shown promise in the early detection of infection and systemic inflammation.

Approximately 100 patients aged 65 years or older who are admitted to the hospital with a low-energy hip fracture will be included in this study. Blood tests will be performed at hospital admission, after surgery, and at other time points as part of standard clinical care. These tests include routine blood counts and inflammatory markers such as C-reactive protein (CRP), procalcitonin (PCT), antithrombin III, and MDW. No additional invasive procedures are required beyond standard medical care.

Researchers will collect information about each patient's medical history, overall health status, and daily activity level before the fracture. Patients will be followed after surgery to assess complications, length of hospital stay, and survival at 1 month, 3 months, and 1 year.

The results of this study may help determine whether MDW can be used as a simple and reliable marker to identify patients at higher risk of complications or death after hip fracture. This could support earlier intervention, closer monitoring, and improved care for elderly patients with hip fractures in the future.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥65 years
* Admission with low-energy hip fracture (femoral neck, intertrochanteric, or subtrochanteric fracture)
* Admission to General Hospital of Attica KAT
* Availability of baseline laboratory measurements, including complete blood count with monocyte distribution width (MDW) and inflammatory biomarkers

Exclusion Criteria:

* Age <65 years
* High-energy trauma-related hip fractures
* Pathological fractures

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The study population includes approximately 100 geriatric patients aged 65 years and older admitted with low-energy hip fractures and treated surgically at the 2nd Orthopaedic Department of the General Hospital of Attica KAT. Participants undergo routine perioperative evaluation, including demographic and clinical data collection and laboratory assessment of inflammatory biomarkers such as monocyte distribution width (MDW), C-reactive protein, procalcitonin, and antithrombin III. Patients are followed prospectively to evaluate postoperative morbidity and all-cause mortality at 1 month, 3 months, and 12 months following surgery.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | Up to 12 months postoperatively.
  Assessment of all-cause mortality in geriatric patients with low-energy hip fracture and its association with Monocyte Distribution Width (MDW) values measured at admission and during hospitalization.

SECONDARY OUTCOMES:
Postoperative morbidity | From postoperative day 1 through study completion, an average of 1 year.
  Assessment of postoperative morbidity, including infectious and non-infectious complications, and its association with Monocyte Distribution Width (MDW) and other inflammatory markers (C-reactive protein, procalcitonin, antithrombin III).
Incidence of sepsis | From postoperative day 1 through study completion, an average of 1 year.
  Occurrence of sepsis during hospitalization or postoperative follow-up, evaluated in relation to MDW values and other inflammatory biomarkers.
Change in Monocyte Distribution Width (MDW) over time | From hospital admission through hospital discharge, up to 14 days postoperatively.
  Evaluation of changes in MDW values from admission through the postoperative period and at discharge, and their association with clinical outcomes.
Length of hospital stay | From the date of hospital admission until hospital discharge, assessed up to 30 days.
  Duration of hospitalization measured in days and its association with MDW and inflammatory marker levels.

CONTACTS AND LOCATIONS:
Overall Officials: Efstathios Chronopoulos, Study Director — KAT General Hospital, Athens Greece
Locations (1):
- Laboratory for Research of the Musculoskeletal System, Kifissia, Attica, Greece

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will be made available to qualified researchers upon reasonable request. Data sharing will comply with the General Data Protection Regulation (EU GDPR) and applicable ethical and institutional requirements. Requests must include a brief description of the intended research use. Approved requests will be granted access to fully anonymized data sets, ensuring that study participants cannot be identified.